CLINICAL TRIAL: NCT04957992
Title: Infant Formula and Toddler Drink Feeding Intervention Through 24 Months of Age
Brief Title: BIG Study (Brain, Immune, and Gut Health Evaluation of Infants/Young Children Fed Infant Formula, and Later Supplemental Toddler Nutrition, With 5 Specific HMOs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL51
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Growth
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Feeding Group (Active Comparator): Milk based product
  Interventions: Other: Control Infant Formula; Other: Control Toddler Drink
- Experimental Feeding Group (Experimental): Milk based product with oligosaccharides
  Interventions: Other: Experimental Infant Formula; Other: Experimental Toddler Drink
- Human Milk Reference Group (Other): Human Milk
  Interventions: Other: Human Milk; Other: Human Milk Supplemental Formula; Other: Human Milk Toddler Drink

INTERVENTIONS:
Other: Control Infant Formula — Ad libitum or as instructed by HCP, feeding period from enrollment to 12 months of age
  Arms: Control Feeding Group
Other: Control Toddler Drink — ~ 16 fl oz per day as primary milk beverage; feeding period from 12 to 24 months of age
  Arms: Control Feeding Group
Other: Experimental Infant Formula — Ad libitum or as instructed by HCP, feeding period from enrollment to 12 months of age
  Arms: Experimental Feeding Group
Other: Experimental Toddler Drink — ~ 16 fl oz per day as primary milk beverage; feeding period from 12 to 24 months of age
  Arms: Experimental Feeding Group
Other: Human Milk — Ad libitum or as instructed by HCP
  Arms: Human Milk Reference Group
Other: Human Milk Supplemental Formula — Ad libitum if consuming supplemented formula; feeding period up to 12 months of age
  Arms: Human Milk Reference Group
Other: Human Milk Toddler Drink — ~16 fl oz per day if providing supplemental nutrition other than HM; feeding period from 12 to 24 months of age
  Arms: Human Milk Reference Group

SUMMARY:
The purpose of this study is to evaluate the growth and development outcomes of infants fed a new infant formula and toddler drink through 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good health as determined from participant's medical history
* Participant is a singleton from a full-term birth with a gestational age of 37 - 42 weeks by parent report
* Participant's birth weight was ≥ 2490 g (~5 lbs. 8 oz.)
* Parent(s) confirm their intention to feed their infant the study product as the sole source of feeding from Study Visit 1 to 6 months of age, and as the sole milk beverage during the first 12 months of life
* Parent(s) confirm their intention to feed the infant the assigned toddler drink from 12 months of life to 24 months of life as the primary milk beverage
* Parent(s) confirm their intention not to administer vitamin or mineral supplements,(except for vitamin D supplements if instructed by their healthcare professional) from enrollment through the duration of the study
* Parent(s) confirm their intention not to administer solid foods or juices to the infant from enrollment through 6 months of age unless recommended by the participant's HCP
* Participant's parent(s) has voluntarily signed and dated an informed consent form (ICF), approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study
* If parent(s) elect to feed the participant human milk, they confirm that their infant was fed human milk since birth and confirm their intention to exclusively feed human milk as the sole source of feeding through 6 months of age.
* If parent(s) of human milk fed participant elect to supplement or wean, they confirm their intention to use the experimental supplemental/weaning formula and experimental toddler drink as the primary milk beverage.

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development
* Awareness of a positive drug screen (including but not limited to cocaine, heroin, or methamphetamine) in the mother or participant
* Suspected maternal substance abuse including alcohol
* Participant is taking and plans to continue medications (including over the counter (OTC), such as Mylicon® for gas), home remedies (such as juice for constipation), herbal preparations, prebiotics or probiotics, or rehydration fluids that might affect GI tolerance
* Participant is in another study that has not been approved as a concomitant study by AN
* Participant has been treated with antibiotics (except for topical antibiotics, eye drops) prior to enrollment
* Participant has been treated with other medications (besides antibiotics) that in the opinion of the PI may affect growth, GI tolerance and/or development, prior to enrollment

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 607 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Growth | Study Day 1 to 6 Months of Age
  weight for age z-score

SECONDARY OUTCOMES:
Incidence of respiratory infection between study groups | Study Day 1 to 24 Months of Age
  Adverse event reports
Number of respiratory infection episodes between study groups | Study Day 1 to 24 Months of Age
  Adverse event reports
Incidence of infection morbidity between study groups | Study Day 1 to 24 Months of Age
  Adverse event reports
Number of episodes of infection morbidity between study groups | Study Day 1 to 24 Months of Age
  Adverse event reports
Weight | Study Day 1 to 24 Months of Age
  Interval weight gain per day
Length | Study Day 1 to 24 Months of Age
  Interval length gain per day
Head Circumference | Study Day 1 to 24 Months of Age
  Interval head circumference gain per day
Gastrointestinal Tolerance | Study Day 1 to 12 months of Age
  Parent completed diary

OTHER OUTCOMES:
Formula Satisfaction Questionnaire | 28 Days of Age to 6 Months of Age
  Parent completed questionnaire; 12 questions with 5-point Likert scale questions scaled from positive to negative
Toddler Drink Satisfaction Questionnaire | 18 Months of Age to 24 Months of Age
  Parent completed questionnaire; 12 questions with 5-point Likert scale questions scaled from positive to negative
Infant Feeding and Stool Patterns Questionnaire | 28 Days of Age to 119 Days of Age]
  Parent completed questionnaire; 16, 5-point Likert scale questions, scaled from Always to Never
Infant and Toddler Behavior Questionnaire | 119 Days of Age
  Parent completed questionnaire; 22 questions with 5-point Likert scale questions, scaled from Always to Never
Product Intake | Study Day 1 to 24 Months of Age
  Parent completed intake diary
Dietary Intake | 6 Months of Age to 24 Months of Age
  Parent completed 24-hour recall
Stool Sample | Study Day 1 to 24 Months of Age
  Microbiota characterization; Subset of subjects
Bayley™-4 Scale of Infant & Toddler Development IV | 12 Months of Age to 24 Months of Age
  Examiner rated assessment; Scores are totaled and compared to normative age group data and between groups; Subset of subjects
MacArthur Communicative Developmental Inventory (CDI)/Words and Gestures and CDI)/Words and Sentences | 12 Months of Age to 24 Months of Age
  Parent completed questionnaire of Words and Gestures and Words and Sentences; Percentiles compared to normative group data and between groups
Modified Home Short Form | 6 Months of Age to 24 Months of Age]
  Parent completed questionnaire; 8 questions related to the home environment adapted from the HSF compared between groups
Medications | Study Day 1 to 24 Months of Age
  Medication usage including frequency and reason for use
Adverse Events | Study Day 1 to 24 Months of Age
  Parent reported adverse events
Health Resource Utilization | Study Day 1 to 24 Months of Age
  Number of visits
Missed Parental Work Days | Study Day 1 to 24 Months of Age
  Parent reported number of days
Blood Collection | 6 and 24 Months of Age
  Blood Immune Markers; Subset of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reverri, PhD, MS, RD, Study Chair — Abbott Nutrition
Locations (42):
- United States (42):
  - MedPharmics, LLC 3192, Phoenix, Arizona
  - HealthStar Research, Glenwood, Arkansas
  - HealthStar Research, LLC, Hot Springs, Arkansas
  - The Children's Clinic of Jonesboro, P.A., Jonesboro, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Optumcare Colorado Springs, LLC, Colorado Springs, Colorado
  - Boeson Research 3266, Grand Junction, Colorado
  - TOPAZ Clinical Research, Inc., Apopka, Florida
  - Columbus Clinical Services, LLC., Miami, Florida
  - Emerald Coast OBGYN Clinical Research, Panama City, Florida
  - ASCLEPES Research Centers, Spring Hill, Florida
  - Jedidiah Clinical Research, Tampa, Florida
  - Meridian Clinical Research 3259, Macon, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Leavitt Clinical Research, Idaho Falls, Idaho
  - Qualmedica Research, Evansville, Indiana
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - MedPharmics, LLC 3343, Covington, Louisiana
  - MedPharmics Research 3369, Slidell, Louisiana
  - Boeson Research 3367, Great Falls, Montana
  - Boeson Research 3265, Kalispell, Montana
  - Boeson Research 3267, Missoula, Montana
  - Meridian Clinical Research 3264, Grand Island, Nebraska
  - Meridian Clinical Research 3263, Hastings, Nebraska
  - Meridian Clinical Research 3304, Lincoln, Nebraska
  - Alivation Research, Lincoln, Nebraska
  - University of Nebraska Medical Center 3315, Omaha, Nebraska
  - University of Nebraska Medical Center 3314, Omaha, Nebraska
  - Advantage Clinical Trials, The Bronx, New York
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Tribe Clinical Research LLC 3313, Greenville, South Carolina
  - Tribe Clinical Research LLC 3382, Spartanburg, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Holston Medical Group 3301, Bristol, Tennessee
  - Holston Medical Group 3046, Kingsport, Tennessee
  - AVIATI Healthcare & Clinical Research, Memphis, Tennessee
  - Javara Inc. 3377, Dallas, Texas
  - Maximos Ob/Gyn, League City, Texas
  - National Clinical Research, Inc, Richmond, Virginia
  - Multicare Health System - Rockwood Pediatrics, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No